CLINICAL TRIAL: NCT03942172
Title: Treatment of Balance Disorders in Parkinson's Patients Using SpotOn Balance Glasses
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study protocol needed to be modified
Sponsor: SpotOn Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SpotOn_03
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpotOn Balance (Experimental): SpotOn Balance Glasses
  Interventions: Device: SpotOn balance glasses

INTERVENTIONS:
Device: SpotOn balance glasses — SpotOn Balance Glasses comprising of personalized visual stimuli placed on the glasses's lenses

SUMMARY:
An open-label study to evaluate the effect of SpotOn balance glasses in non-demented Parkinson's patients with balance disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Female or men
2. Diagnosed with Parkinson's disease (according to Brain Bank UK criteria)
3. Non-demented
4. Age: ≥ 30 years
5. Gait disturbances
6. Patients who are able to perform questionnaires and physical tests (including computerized tests)
7. Gave informed consent for participation in the study

Exclusion Criteria:

1. Unstable (less than 1 month) use of concomitant medications that might affect the balance system
2. Change of PD medications during the past month
3. Any medical condition or disorder that could produce gait or balance disturbances unless well controlled for at least 3 months
4. Blindness
5. Currently taking part in a clinical trial or within 30 days prior to screening
6. Any known condition which in the opinion of the investigator may impair gait or balance and/or limits the successful trial completion

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's disease rating scale | 3 weeks
  A comprehensive 50 question clinical rating scale for the assessment of both motor and non-motor symptoms associated with Parkinson's. The total cumulative score will range from 0 (no disability) to 199 (total disability).
TIMED UP AND GO (TUG) | 3 weeks
  The TUG test is a physical performance measure in which the ability to rise up from a seated chair position, walk 3m, turn, walk back, and sit down is timed.
Berg Balance Scale (BBS) | 3 weeks
  The BBS is a widely used clinical test of a person's static and dynamic balance abilities. t is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.A score of 56 indicates functional balance.
Non-Motor Symptoms Scale (NMSS) | 3 weeks
  The non-motor symptoms questionnaire is a 30-point, patient-based questionnaire used to determine the non-motor symptoms experienced by the patient during the past month.Responses quantify symptoms according severity (using a scale of 0-3) and frequency (using a scale of 0-4). Higher scores represent more severe and more frequent symptoms.
39-item Parkinson's Disease Questionnaire (PDQ-39) | 3 weeks
  This questionnaire assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. It is scored on a scale of 0-100, with lower scores indicating better health and high scores more severe symptoms.
Freeze of gait (FOG) Questionnaire | 3 weeks
  Consists of 16 items assessing freeze of gait. Total score ranges from 0 to 24, higher score corresponds to more severe FOG.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Shlezinger, MD, Principal Investigator — Rambam Hospital
Locations (1):
- RAMBAM Health centre, Haifa, Israel